CLINICAL TRIAL: NCT04314531
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Demonstrate the Efficacy and Safety of Tildrakizumab in Anti-TNF Naïve Subjects With Active Psoriatic Arthritis II (INSPIRE 2)
Brief Title: Efficacy and Safety of Tildrakizumab Compared to Placebo in Anti-TNF naïve Subjects With Active Psoriatic Arthritis II (INSPIRE 2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TILD-19-19
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Active Psoriatic Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: TILD
- Arm B (Placebo Comparator)
  Interventions: Drug: matching placebo injections

INTERVENTIONS:
Drug: TILD — one 1 mL injection of study medication
  Arms: Arm A
Drug: matching placebo injections — one 1 mL injection of placebo
  Arms: Arm B

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, Phase 3 study to evaluate the efficacy and safety of tildrakizumab compared to placebo in anti-TNF naïve subjects with active PsA .

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent.
2. Subject is ≥ 18 years of age at time of Screening.
3. Subject has a diagnosis of active PsA for at least 6 months before the first administration of the study agent and has active PsA at Screening or Baseline.
4. Rheumatoid factor (RF) and anti-cyclic citrullinated peptide antibodies (anti-CCP Ab) negative.
5. Subjects must have no prior exposure to anti-tumor necrosis factor (anti-TNF) agent(s) use for the treatment of PsO or PsA.

Exclusion Criteria:

1. The subject has a planned surgical intervention between Baseline and the Week 52 evaluation for a pretreatment condition.
2. Subject has an active infection or history of infections as follows:

   * any active infection for which systemic anti-infectives were used within 28 days prior to first IMP dose, with the last dose having been received within 7 days of Screening,
   * a serious infection, defined as requiring hospitalization or intravenous (IV) anti-infectives within 8 weeks prior to the first IMP dose, with the last dose having been received within 7 days of Screening,
   * recurrent or chronic infections, e.g., chronic pyelonephritis, chronic osteomyelitis, bronchiectasis, or other active infection that, in the opinion of the Investigator, might cause this study to be detrimental to the subject.
3. Subject has any concurrent medical condition or uncontrolled, clinically significant systemic disease (e.g., renal failure, heart failure, hypertension, liver disease, diabetes, or anemia) that, in the opinion of the Investigator, could cause this study to be detrimental to the subject.
4. Subject has a known history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
5. Subject had myocardial infarction, unstable angina pectoris, or ischemic stroke within the past 6 months prior to the first IMP dose.
6. Subject has any active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma.
7. Subjects with a history of alcohol or drug abuse in the previous 2 years.
8. Female subjects of childbearing potential who do not agree to abstain from heterosexual activity or practice a dual method of contraception, for example, a combination of the following: (1) oral contraceptive, depo progesterone, or intrauterine device; and (2) a barrier method (condom or diaphragm). Male subjects with female partners of childbearing potential who are not using birth control as described above must use a barrier method of contraception (e.g., condom) if not surgically sterile (i.e., vasectomy). Contraceptive methods must be practiced upon signing the Informed Consent and through 24 weeks after the last dose of IMP. If a subject discontinues prematurely, the contraceptive method must be practiced for 17 weeks following final administration of IMP. A follicle-stimulating hormone (FSH) test should be performed to confirm menopause (per reference values of the laboratory) for those women with no menses for less than 1 year.
9. Subject currently enrolled in another investigational device/procedure or drug study, or Baseline of this study is less than 30 days or 5 half-lives (whichever is longer) since ending another investigational device/procedure or drug study(s), or receiving other investigational agent(s).
10. Subject previously has been enrolled (randomized) in this study.
11. Subject has any kind of disorder that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.
12. Donation or loss of 400 milliliter (mL) or more of blood within 8 weeks before first dose of IMP.
13. Subjects who have been placed in an institution on official or judicial orders.
14. Subjects who are related to or dependent on the Investigator, Sponsor, or study site such that a conflict of interest could arise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieve American College of Rheumatology [ACR20] | at Week 24
  the proportion of subjects achieving a 20% reduction from Baseline in response criteria

SECONDARY OUTCOMES:
The proportion of subjects achieving American College of Rheumatology [ACR50] | at Week 24
  the proportion of subjects achieving a 50% reduction from Baseline in response criteria
The proportion of subjects achieving American College of Rheumatology [ACR70] | at Week 24
  the proportion of subjects achieving a 70% reduction from Baseline in response criteria
The proportion of subjects achieving Psoriasis Area and Severity Index 75 response among subjects with body surface area ≥3% at baseline | at Weeks 24
The change from Baseline in the van der Heijde modified total Sharp score | Week 24
The change from Baseline in the van der Heijde modified total Sharp score | at Week 16
The Change from Baseline in American College of Rheumatology Response Criteria Components Score | at Week 24
  Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Assessment of Arthritis Pain (Visual Analog Scale, 0-100), C-reactive protein levels and erythrocyte sedimentation rate levels
The change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index | at Week 24
The change from Baseline in Leeds Enthesitis Index | at Week 24
The change from Baseline in Leeds Dactylitis Index | at Week 24
The proportion of subjects who achieve a Disease Activity Score-C-reactive protein < 3.2 | at Week 24
The change from Baseline in van der Heijde modified Sharp sub-scores (erosion score and joint space narrowing score) | at Week 24
The proportion of subjects with the Change in van der Heijde modified total Sharp score <0 and < 0.5 | Week 24
The proportion of subjects with active Psoriasis and body surface area ≥3% | at Week 24
  Psoriasis Area and Severity Index 90 and Psoriasis Area and Severity Index 100
The change from Baseline in anti-tumor necrosis factor naïve subjects with active Psoriasis and body surface area ≥ 3% (those with involvement of nails) | at Week 24
  Physician Global Assessment-Psoriasis and nail psoriasis severity index
The proportion of subjects achieving American College of Rheumatology [ACR20, ACR50 and ACR70] | at Week 52
  the proportion of subjects achieving a 20/50/70% reduction from Baseline in response criteria
The change from Baseline in American College of Rheumatology Response Criteria Components Score | at week 52
  Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Assessment of Arthritis Pain (Visual Analog Scale, 0-100), C-reactive protein levels and erythrocyte sedimentation rate levels
change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index | at Week 52
The change from Baseline in Leeds Enthesitis Index, Leeds Dactylitis Index and Health Assessment Questionnaire Disability Index score | at Week 52
The proportion of subjects who achieve a Disease Activity Score(28 [joints]-C-reactive protein) < 3.2 | at Week 52
The change from Baseline in van der Heijde modified total Sharp score | at Week 52
The change from Baseline in van der Heijde modified Sharp sub-scores (erosion score and joint space narrowing score) | at Week 52
The proportion of subjects with the change in van der Heijde modified total Sharp score <0 and < 0.5 | at Week 52
In anti-tumor necrosis factor naïve subjects with active Psoriasis and body surface area ≥3%, the proportion of subjects with Psoriasis Area and Severity Index 75, Psoriasis Area and Severity Index 90 and Psoriasis Area and Severity Index 100 | at Week 52
In anti-tumor necrosis factor naïve subjects with active Psoriasis and body surface area ≥3% those with involvement of nails, the change from Baseline in nail psoriasis severity index | at Week 52
In anti-tumor necrosis factor naïve subjects with active Psoriasis and body surface area ≥3%, the change from Baseline in Physician Global Assessment-Psoriasis | at week 52
Change from baseline in health assessment questionnaire - disability index (HAQ-DI) score | at Week 24
The change from Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components | measured timepoints
The change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scores | at week 24

OTHER OUTCOMES:
The proportion of subjects achieving American College of Rheumatology [ACR20] | exclusive of Weeks 24 and 52
  the proportion of subjects achieving a 20% reduction from Baseline in response criteria
The proportion of subjects achieving American College of Rheumatology [ACR50] | exclusive of Weeks 24 and 52
  the proportion of subjects achieving a 50% reduction from Baseline in response criteria
The proportion of subjects achieving American College of Rheumatology [ACR70] | exclusive of Weeks 24 and 52
  the proportion of subjects achieving a 70% reduction from Baseline in response criteria
he change from Baseline in American College of Rheumatology Response Criteria Components Score | exclusive of Weeks 24 and 52
  Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Assessment of Arthritis Pain (Visual Analog Scale, 0-100), C-reactive protein levels and erythrocyte sedimentation rate levels
The change from Baseline in Leeds Enthesitis Index, Leeds Dactylitis Index, Bath Ankylosing Spondylitis Disease Activity Index and Health Assessment Questionnaire Disability Index score | exclusive of Weeks 24 and 52
The proportion of subjects who achieve a Disease Activity Score-C-reactive protein < 3.2 | exclusive of Weeks 24 and 52
The proportion of subjects with active Psoriasis and body surface area ≥ 3% with Psoriasis Area and Severity Index 75, Psoriasis Area and Severity Index 90 and Psoriasis Area and Severity Index 100 | exclusive of Weeks 24 and 52
The change from Baseline in the levels of "Metabolic Biomarkers" | at Week 24
the change from baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) | at Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 52
proportion of subjects who achieve a response based on Modified Psoriatic Arthritis Responder Criteria (PsARC) | at Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 52.
change from baseline in Work Productivity and Activity Impairment Questionnaire Scores | at Week 12,16 24, 48 and 52.
change from baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) | at Week 8,16, 24 and 52.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (11):
  - Sunpharma site no. 12, Covina, California
  - Sunpharma site no. 04, Miami Beach, Florida
  - Sunpharma site no. 02, New Port Richey, Florida
  - Sunpharma site no. 07, Tamarac, Florida
  - Sunpharma site no. 05, Springfield, Missouri
  - Sunpharma site no. 10, Lincoln, Nebraska
  - Sunpharma site no. 11, Greenville, South Carolina
  - Sunpharma site no. 09, Lubbock, Texas
  - Sunpharma site no. 03, San Antonio, Texas
  - Sunpharma site no. 01, Tomball, Texas
  - Sunpharma site no. 06, Spokane, Washington
- Australia (2):
  - Sunpharma Site 39, Phillip, Australian Capital Territory
  - Sunpharma site no. 08, Hobart, Tasmania
- Czechia (3):
  - Sunpharma Site 64, Brno
  - Sunpharma Site 97, Prague
  - Sunpharma Site 63, Zlín
- Germany (2):
  - Sunpharma Site 73, Berlin
  - Sunpharma Site 92, Herne
- India (8):
  - Sunpharma Site 111, Surat, Gujarat
  - Sunpharma Site 110, Bangalore, Karnataka
  - Sunpharma Site 107, Belagavi, Karnataka
  - Sunpharma Site 109, Hubli, Karnataka
  - Sunpharma Site 108, Pune, Maharashtra
  - Sunpharma Site 112, Hyderabad, Telangana
  - Sunpharma Site 106, Lucknow, Uttar Pradesh
  - Sunpharma Site 113, Kochi
- Japan (11):
  - Sunpharma Site 84, Nagoya, Aichi-ken
  - Sunpharma Site 89, Kitakyushu, Fukuoka
  - Sunpharma Site 86, Sendai, Miyagi
  - Sunpharma Site 24, Miyazaki, Miyazaki
  - Sunpharma Site 91, Mitaka, Tokyo
  - Sunpharma Site 85, Shinjuku, Tokyo
  - Sunpharma Site 90, tabashi City, Tokyo
  - Sunpharma Site 22, Kitakyushu-shi
  - Sunpharma Site 88, Kumamoto
  - Sunpharma Site 87, Osaka
  - Sunpharma Site 23, Tsu
- Poland (5):
  - Sunpharma Site 93, Bialystok
  - Sunpharma Site 95, Bialystok
  - Sunpharma Site 94, Lublin
  - Sunpharma Site 74, Poznan
  - Sunpharma Site 96, Warsaw
- South Korea (3):
  - Sunpharma Site 18, Incheon
  - Sunpharma Site 20, Seoul
  - Sunpharma Site 19, Seoul
- Spain (4):
  - Sunpharma Site 75, A Coruña
  - Sunpharma Site 71, Córdoba
  - Sunpharma Site 100, Madrid
  - Sunpharma Site 72, Seville

IPD SHARING:
Plan to Share IPD: No